CLINICAL TRIAL: NCT06311318
Title: Post-operative Lower Eyelid Massage Versus Standard Care for Prevention of the Lower Eyelid Scare Contracture After Subciliary Approach in Traumatic Facial Fracture Repair, a Randomized Controlled Trial
Brief Title: Post-operative Lower Eyelid Massage for Prevention of the Lower Eyelid Scare Contracture After Subciliary Approach
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Wimon Sirimaharaj, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Department of surgery MED CMU
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Zygomatic and Lefort II Fractures; Infraorbital Rim Fixation; Subciliary Approach Repair
Keywords: subciliary incision; subciliary approach; lower eyelid massage; facial fracture; scar contracture; eyelid malposition; ectropion
MeSH Terms: conditions — Ectropion

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial enrolled patients with traumatic facial fractures slated for subciliary approach repair. Patients were randomly allocated to the lower eyelid massage (experimental) or standard care (control) groups. The massage group received post-operative instructions. Data on demographics, injury profiles, lower eyelid scar contracture (graded by GLESCO criteria), eyelid malpositioning, comfort scores, and complications were gathered over a 6-month follow-up.
Who Masked: Outcomes Assessor
Masking Description: Patients were randomly assigned, using concealed block of four randomization, to either the experimental group receiving lower eyelid massage or the control group receiving standard care. While the authors, acting as massage trainers, were unblinded, an independent plastic surgeon, serving as the assessor, remained blinded to the study interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage group (Experimental): Patients in the experimental group received training and guidance from trained investigators regarding post-operative lower eyelid massage.
  Interventions: Procedure: lower eyelid massage
- Non-massage group (No Intervention): The control group receiving standard care without post-operative lower eyelid massage.

INTERVENTIONS:
Procedure: lower eyelid massage — The massage technique was executed with the patient in a fully open-eyed state, maintaining an upward gaze. The lateral aspect of the distal phalanx of the index finger was employed, exerting pressure on the lower eyelid to bring its margin into contact with the upper eyelid margin for a duration of 10 seconds per repetition. This procedure comprised 10 repetitions per set, administered once hourly, spanning 10 hours daily. The massage instruction was provided either by the authors or plastic surgery residents.
  Arms: Massage group

SUMMARY:
Patients were randomly allocated to the lower eyelid massage (experimental) or standard care (control) groups. The massage group received post-operative instructions. Data on demographics, injury profiles, lower eyelid scar contracture (graded by GLESCO criteria), eyelid malpositioning, comfort scores, and complications were gathered over a 6-month follow-up.

DETAILED DESCRIPTION:
* The massage technique was executed with the patient in a fully open-eyed state, maintaining an upward gaze. The lateral aspect of the distal phalanx of the index finger was employed, exerting pressure on the lower eyelid to bring its margin into contact with the upper eyelid margin for a duration of 10 seconds per repetition. This procedure comprises 10 repetitions per set, administered once hourly, spanning 10 hours daily. The massage instruction was provided either by the authors or plastic surgery residents.
* Facial fracture surgeries were conducted by experienced plastic surgeons and/or proficient 4th and 5th year plastic surgery residents at Chiang Mai University Hospital, utilizing the skin-muscle flap subciliary approach. All patients underwent surgery one week after injury to mitigate soft tissue swelling, which had subsided by that time.
* Consistent pre-operative, peri-operative, and post-operative care protocols were administered to both patient groups. Stitches at the subciliary incision site were extracted on post-operative day 5. Patients in the massage group were instructed to commence lower eyelid massage on the day when stitches were removed.
* The follow-up assessments were occurred at 1-week, 3-week, 6-week, 3-month, and 6-month intervals post-operatively. Evaluation criteria include the Grading of Lower Eyelid Scar Contracture (GLESCO). Additionally, grading of lower eyelid malpositioning, comfort scores, rate on a scale of 0-10, adapted from POSAS and Verbal Rating Scale, wound infection, dehiscence, eyelid comfort, and management related to the subciliary incision will be assessed and documented by the plastic surgeon (author) and plastic surgery resident.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with zygomatic and Lefort II fractures necessitating infraorbital rim fixation following motorcycle accidents, and presenting without external lower eyelid wounds.

Exclusion Criteria:

* Pre-existing lower eyelid retraction (from previous scar, neurogenic cause, myogenic cause or Graves' disease), incision alteration, communication barriers, inability to perform daily activities or lower eyelid massage (ECOG ≥ 2, PPS Adult Suandok ≤ 60), inability to attend follow-up visits, and patient refusal.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Grading of Lower Eyelid Scar Contracture (GLESCO) | The follow-up assessments occurred at 1-week, 3-week, 6-week, 3-month, and 6-month intervals post-operatively.
  An anatomical score adapted by the authors, which was not independently validated as it relies on consistent anatomy across patients.
  Patient in normal neutral gaze, examiner use a finger to push the patient's lower eyelid up to reach upper eyelid, evaluate the lower lid margin compare with cornea Grade 0: Can push lower eyelid up to 100% of cornea Grade 1: Can push lower eyelid up to 75% of cornea Grade 2: Can push lower eyelid up to 50% of cornea Grade 3: Can push lower eyelid up to 25% of cornea Grade 4: Can push lower eyelid less than 25% of cornea
Grading of lower eyelid malpositioning | The follow-up assessments occurred at 1-week, 3-week, 6-week, 3-month, and 6-month intervals post-operatively.
  One of the complications encountered following lower-lid blepharoplasty, ranging in severity from mild lower-lid retraction to frank ectropion with marked lower-lid eversion.
  Patient in normal neutral gaze, examiner observe position and characteristic of lower eyelid.
  Grade 0: Normal eye position Grade 1: Lateral rounding of the eye Grade 2: Central sclera show involving limbus Grade 3: Mild eversion of lower lid with tear pooling in inferior cul-de-sac Grade 4: Frank outward eversion of lower lid with exposure of palpebral conjunctiva
Comfort scores | The follow-up assessments occurred at 1-week, 3-week, 6-week, 3-month, and 6-month intervals post-operatively.
  Represent subjective clinical evaluations by patients, assessing the overall comfort of the eye, including factors like dryness and tightness of the eyelid, rated on a scale of 0-10, adapted from POSAS and Verbal Rating Scale

IPD SHARING:
Plan to Share IPD: No